CLINICAL TRIAL: NCT04288765
Title: Carfilzomib, Daratumumab, Lenalidomide and Dexamethasone as First Line Treatment in Multiple Myeloma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: incomplete recruitment
Sponsor: Grupo Cooperativo de Hemopatías Malignas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAL 319/2019
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Multiple Myeloma
Keywords: Newly diagnosed
MeSH Terms: conditions — Multiple Myeloma | interventions — Injections; Lenalidomide; carfilzomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients with newly diagnosed and previously untreated multiple myeloma living in Mexico that are fit for a quadruple therapy for multiple myeloma. Those patients that aren't fit or unavailable for transplant will go to the continuous treatment arm. The stratification of the study will be done by age and by cytogenetic risk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Non transplant (Experimental): Carfilzomib Lenalidomide Daratumumab Dexamethasone
  Interventions: Drug: Daratumumab Only Product in Parenteral Dose Form
- Group B - transplant (Active Comparator): Carfilzomib Lenalidomide Daratumumab Dexamethasone Autologous stem cell transplantation (ASCT)
  Interventions: Drug: Daratumumab Only Product in Parenteral Dose Form

INTERVENTIONS:
Drug: Daratumumab Only Product in Parenteral Dose Form — Induction = 8 cycles Carfilzomib on Day 1st, 8th and 15th Lenalidomide: Day 1 to 21
  Daratumumab:
  Cycles 1-2: weekly Cycles 3-4: every two weeks Cycles 5-8: every month Dexamethasone: 40 mg weekly
  Other Names: Lenalidomide; Carfilzomib; Dexamethasone

SUMMARY:
Carfilzomib in combination with lenalidomide, daratumumab and dexamethasone (KRDd) can induce profound clinical responses. The investigators want to observe the effectiveness of the quadruple therapy of carfilzomib, lenalidomide, daratumumab and dexamethasone on patients receiving 8 cycles of KRDd with autologous stem cell transplantation versus patients with 8 cycles of KRDd without autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed and previously untreated multiple myeloma by the International Myeloma Working Group criteria that requires treatment based on: Presence of elevated calcium, renal failure, anemia and/or bone lesions (CRAB) Clonal bone marrow plasma cells ³ 60% Involved/uninvolved serum free light chain ratio ³ 100 >1 focal lesions on MRI studies (³5 mm in size)
2. Age > 18 years
3. Functional stage of 0 - 1 measured by the Eastern Cooperative Oncology Group (ECOG) scale.
4. Capacity and willingness to provide a written informed consent.

Exclusion Criteria:

1. POEMS syndrome
2. Systemic amyloidosis
3. Plasma cells leukemia
4. Radiotherapy on multiple sites on the period of 4 weeks before the initiation of treatment (1 week if it is one region)
5. Improper liver function: total bilirubin > 1.5 x upper limit of normal (ULN) or > 3 x ULN in patients with Gilbert syndrome, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 3.0 x ULN.
6. Non-controlled systematic active infection (viral, bacterial and/or fungic).
7. Patients with known infection by human immunodeficiency virus (HIV).
8. Active infection by hepatitis B.
9. Active infection by hepatitis C.
10. Significant cardiovascular diseases as uncontrolled or symptomatic arrhythmias, congestive heart failure or acute myocardial infarction within 2 months prior to screening, or any New York Heart Association (NYHA) class 3 or 4 heart disease.
11. Diagnosis of previous malignancies for 2 years, with exception of patients with basal or squamous cell carcinoma or "in situ" carcinoma of cervix or breast.
12. History of allergic reaction or severe anaphylaxis to humanized or murine monoclonal antibodies.
13. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Complete response with negative minimal residual disease | 10 months
  Complete response with MRD-negative disease measured by inmunophenotype with the International Myeloma Working Group response criteria

SECONDARY OUTCOMES:
Overall survival | 36 months
  Overall survival measured on months on both study groups
Progression free survival | 36 months
  Progression free survival measured on months from the time to the end of treatment to disease progression on both study groups
Rate of Adverse Events | 36 months
  Rate of adverse events rated grade ≥3 by CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo Cooperativo de Hemopatías Malignas, Huixquilucan, State of Mexico, Mexico